CLINICAL TRIAL: NCT04274244
Title: Comparison of Clinical and Radiographic Parameters in the Application of Cross-linked Hyaluronic Acid 1.8% (Hyadent BG®) and Enamel Matrix Derivative (Emdogain®) in Periodontal Regeneration: A Randomized Clinical Trial
Brief Title: Comparison of Clinical and Radiographic Parameters in the Application of Cross-linked Hyaluronic Acid 1.8% and Enamel Matrix Derivative in Periodontal Regeneration.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Valencia (Other)
Collaborators: Regedent AG, Zürich (Unknown)
Responsible Party: Principal Investigator, Andres Lopez Roldan, Associate professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UV3
Record Dates: First submitted 2019-04-09; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Chronic Periodontitis; Periodontal Bone Loss
Keywords: Periodontitis; Hyaluronic acid; Periodontal regeneration
MeSH Terms: conditions — Chronic Periodontitis; Alveolar Bone Loss; Periodontitis | interventions — enamel matrix proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blinding: The researchers who performed the measurements will be different from those who performed the surgery; therefore, the examiner will be blinded during the entire duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cross-Linked Hyaluronate Gel Prefilled Syringe 30 MG/3ML (Experimental): 1. The study participants will first undergo SCALE AND ROOT PLANING. This procedure is the same as that used in the active comparator group and the control group.
  2. Eight weeks following the initial therapy, reevaluation of the intrabony defects in the interproximal sites with a clinical probing depth >5 mm will be performed by radiographs as well as by using William's graduated periodontal probe to confirm the indication for periodontal surgery. Pairs of premolar and molar teeth in the maxilla or the mandible will be randomized to receive the test treatment (REGENERATIVE PERIODONTAL SURGERY with adjunctive hyaluronic acid gel application) or to serve as active comparators (regenerative periodontal surgery with adjunctive enamel matrix derivative application).
  Interventions: Drug: Cross-Linked Hyaluronate Gel Prefilled Syringe 30 MG/3ML
- Enamel Matrix Proteins (Active Comparator): 1. SCALE AND ROOT PLANING
  2. REGENERATIVE PERIODONTAL SURGERY: Application of enamel matrix derivative.
  Interventions: Drug: Enamel Matrix Proteins (Active comparator group)
- Scale and root planning (No Intervention): Control group: Just SCALE AND ROOT PLANING is performed

INTERVENTIONS:
Drug: Cross-Linked Hyaluronate Gel Prefilled Syringe 30 MG/3ML — Regenerative periodontal therapy + Cross-linked hyaluronic acid 1.8%:
  * The modified minimal invasive surgical technique, described by Cortellini 2011, will be used to raise the interdental papilla over the bone defect.
  * Measurement of bone defect with a 0.5mm periodontal probe (PCP-UNC 15, Hu-Friedy Manufacturing, Illinois, USA) to characterize the defect anatomy.
  * Inflammatory tissue will be debrided and the root carefully planed using Gracey curettes.
  * The site will be washed with physiologic sterile solution, dried and the root wil be conditioned with 24% Ethylenediamine tetraacetic acid (EDTA) for two minutes, then the defect area will be carefully rinsed with sterile saline to remove any residual EDTA.
  * Application of Hyadent BG® 1,8% filling the bone defect from the bottom upwards in the test group.
  * Single internal modified mattress suture (5/0 Vicryl, Ethicon).
  * Sutures will be removed after two weeks.
  Other Names: REGENERATIVE PERIODONTAL SURGERY (Test group)
  Arms: Cross-Linked Hyaluronate Gel Prefilled Syringe 30 MG/3ML
Drug: Enamel Matrix Proteins (Active comparator group) — Regenerative periodontal therapy + Enamel matrix proteins:
  * The modified minimal invasive surgical technique, described by Cortellini 2011, will be used to raise the interdental papilla over the bone defect.
  * Measurement of bone defect with a 0.5mm periodontal probe (PCP-UNC 15, Hu-Friedy Manufacturing, Illinois, USA) to characterize the defect anatomy.
  * Inflammatory tissue will be debrided and the root carefully planed using Gracey curettes.
  * The site will be washed with physiologic sterile solution, dried and the root wil be conditioned with 24% Ethylenediamine tetraacetic acid (EDTA) for two minutes, then the defect area will be carefully rinsed with sterile saline to remove any residual EDTA.
  * Application of Emdogain® filling the bone defect from the bottom upwards in the active comparator group.
  * Single internal modified mattress suture (5/0 Vicryl, Ethicon).
  * Sutures will be removed after two weeks.
  Other Names: REGENERATIVE PERIODONTAL SURGERY
  Arms: Enamel Matrix Proteins

SUMMARY:
The aim of this study is to compare the effectiveness in periodontal regeneration of cross-linked hyaluronic acid at 1.8% (Hyadent BG®) with enamel matrix derivative (Emdogain®) in periodontal bone defects evaluating their clinical and radiographic variables.

DETAILED DESCRIPTION:
A high molecular weight polysaccharide, hyaluronic acid, also known as hyaluronan or hyaluronate, has recently been studied as a promising mediator for periodontal regeneration. It has a significant role in mineralized and non-mineralized periodontal tissues for the functioning of its extracellular matrices. It has a multifunctional role in periodontics including the stimulation of cell migration, proliferation and differentiation and the acceleration of wound healing by stimulating angiogenesis. It is used in surgical procedures due to its osteoinductive potential. HA is a key element in soft periodontal tissues, the gingiva and periodontal ligament, and in hard tissue, such as alveolar bone and cementum. It has many structural and physiological functions within these tissues.

This research proposes two experimental groups to whom one of them will be applied cross-linked hyaluronic acid at 1.8% and another group with enamel matrix derivative, and a control group.

The investigator's hypothesis is that the hyaluronic acid shows potential for periodontal regeneration when evaluating its clinical and radiographic variables and when compared with the use of Enamel matrix derivative.

ELIGIBILITY:
Inclusion Criteria:

1. Periodontitis stage II or III, grade A or B: based on the "Consensus report of workgroup of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions" Tonetti 2017. Clinical attachment loss of 3-5mm, radiographic bone loss to the middle third, loss of teeth ≤4 due to periodontitis, probing depth ≥ 6 mm.
2. At least, 20 teeth in the mouth.
3. Plaque Index (PI) < 1, following initial nonsurgical periodontal therapy and hygiene instructions.
4. At least one interproximal 2, 3-wall bone defect with moderate to deep intrabony defects (≥3mm) on the radiographs, and clinical probing depths (PD) >5mm using William's graduated periodontal probe on premolars or molars following initial nonsurgical periodontal therapy.
5. Absence of caries or overflowing restorations and periapical injuries of the target tooth.
6. Non-smokers.
7. Absence of systemic disease.
8. Negative history for pregnancy
9. No relevant medical history that contraindicate periodontal surgery.
10. All participants signed an inform consent form.
11. The participant is female or male adult of ≥ 18 years. The sample in sex will be compensated.
12. The participant is willing and able to return to the treatments and evaluations programmed throughout this clinical study.

Exclusion Criteria:

1. The participant is pregnant or lactating or plans to become pregnant within the next 6 months.
2. Heavy smoker (>10 cigarettes/day).
3. The participant takes> 4 U of alcohol / day.
4. The participant has a chronic illness or decreased mental capacity which would mitigate the ability to comply with the protocol.
5. Taking drugs that could alter the participant's response in healing or with oral concomitant manifestations that, in the opinion of the investigator, could interfere with the assessment of safety or efficacy.
6. Participants with systemic diseases that interfere with treatment such as, Diabetes mellitus, or rheumatoid arthritis.
7. Allergies to drug compounds.
8. The participant has been treated with antibiotics within 3 months before starting the study or has any other systemic condition that requires antibiotic coverage for routine periodontal procedures (eg, heart disease, prosthetic joints, etc.).
9. Participants should not have received periodontal tretment within the 6-month period prior to study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Clinical measure: Clinical attachment loss (CAL). Changes will be assessed at 3 time points. | 1. Baseline, 2. Reevaluation (60 days after root debridement), 3. Second reevaluation (180 days after Periodontal regenerative surgery).
  It is defined as the distance in millimeters between CEJ and the end of the periodontal pocket. The calculation of the depth of the pocket + gingival recession or pocket depth - gingival hyperplasia will be carried out.

SECONDARY OUTCOMES:
Radiographic measure: Cemento-enamel junction (A1) | 1. Baseline, 2. Second reevaluation (180 days after Periodontal regenerative surgery).
  • The cemento-enamel junction (CEJ)of the tooth involved in the intrabony defect.
Radiographic measure: B1 | 1. Baseline, 2. Second reevaluation (180 days after Periodontal regenerative surgery).
  The most coronal position of the alveolar bone crest of the intrabony defect when it touches the root surface of the adjacent tooth before treatment (the top of the crest).
Radiographic measure: D1 | 1. Baseline, 2. Second reevaluation (180 days after Periodontal regenerative surgery).
  The most apical extension of the intrabony destruction where the periodontal ligament space still retained its normal width before treatment (the bottom of the defect).
Clinical measure: Probing pocket depth (PPD). Changes will be assessed at 3 time points. | 1. Baseline, 2. Reevaluation (60 days after Scale and root planing), 3. Second reevaluation (180 days after Periodontal regenerative surgery).
  The probing depth will be measured in six areas (disto-buccal, mediate-vestibular, mesio-buccal, disto-palatal, mid-palatal, and mesio-palatal) of each tooth with a Williams PQ-OW 208 396 probe. It will be use with a pressure of 20 grams that is equivalent to the pressure of dropping the weight of the probe without exerting additional pressure.
Clinical measure: Gingival recession (GR). Changes will be assessed at 3 time points. | 1. Baseline, 2. Reevaluation (60 days after Scale and root planing), 3. Second reevaluation (180 days after Periodontal regenerative surgery).
  The "Full mouth bleeding score" (FMBS) will be calculated based on scores of 0 (no bleeding) or 1 (bleeding) after probing depths are checked. The usual thing is to measure 4 points for each tooth, but we have modified the index and we value 6 points per tooth (disto-buccal, mid-buccal, mesio-buccal, disto-palatal, mid-palatal and mesio-palatal).
  We consider that the score is 1 when we see a red dot in the% bleeding diagram of the periodontogram and 0 when we see the blank box.
Clinical measure: Tooth mobility (TM) Miller (1950). Changes will be assessed at 3 time points. | 1. Baseline, 2. Reevaluation (60 days after Scale and root planing), 3. Second reevaluation (180 days after Periodontal regenerative surgery).
  * Class I: Mobility up to 1 mm in the horizontal direction.
  * Class II: Mobility greater than 1 mm in the horizontal direction.
  * Class III: Excessive movement in both horizontal and vertical directions.
Clinical measure: Furcation involvement: Hamp (1975). Changes will be assessed at 3 time points. | 1. Baseline, 2. Reevaluation (60 days after Scale and root planing), 3. Second reevaluation (180 days after Periodontal regenerative surgery).
  The plaque will be quantified as follows:
  * Score 0 = no plaque
  * Score 1 = A film of plaque adhered to the free gingival margin and the adjacent area of the tooth. The plaque can be seen in situ only after the application of a plaque revealer or by using the probe on the surface of the tooth.
  * Score 2 = moderate accumulation of soft deposits in the pocket, tooth or gingival margin, which can be seen with our eyes.
  * Puntuación 3 = Abundance of soft material inside the bag and / or on the tooth and the gingival margin.
  The evaluation will be carried out in 4 points per tooth (disto-buccal, mesio-buccal, disto-palatal, mesio-palatal).
Clinical measure: Plaque Index (Sillness y Löe 1964). Changes will be assessed at 3 time points. | 1. Baseline, 2. Reevaluation (60 days after Scale and root planing), 3. Second reevaluation (180 days after Periodontal regenerative surgery).
  The plaque will be quantified as follows:
  * Score 0 = no plaque
  * Score 1 = A film of plaque adhered to the free gingival margin and the adjacent area of the tooth. The plaque can be seen in situ only after the application of a plaque revealer or by using the probe on the surface of the tooth.
  * Score 2 = moderate accumulation of soft deposits in the pocket, tooth or gingival margin, which can be seen with our eyes.
  * Puntuación 3 = Abundance of soft material inside the bag and / or on the tooth and the gingival margin.
  The evaluation will be carried out in 4 points per tooth (disto-buccal, mesio-buccal, disto-palatal, mesio-palatal).

CONTACTS AND LOCATIONS:
Overall Officials: Andrés López Roldán, Study Director — University of Valencia; Manuel Rodríguez Aranda, Principal Investigator — University of Valencia; Francisco Alpiste Illueca, Study Director — University of Valencia

REFERENCES:
- [Derived] Rodriguez-A M, Montiel-Company JM, Alpiste-Illueca F, Rodriguez-A L, Paredes-Gallardo V, Lopez-Roldan A. Comparision of crosslinked hyaluronic acid vs. enamel matrix derivative for periodontal regeneration: an 18-month follow-up randomized clinical trial. Clin Oral Investig. 2025 Mar 19;29(4):197. doi: 10.1007/s00784-025-06278-5. PMID 40106008